CLINICAL TRIAL: NCT02040818
Title: RCT for the Treatment of Hemodialysis Catheter-Related Bacteremia
Brief Title: Treatment of Hemodialysis Catheter-Related Bacteremia
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: no enrollment
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Saima Aslam, Adj Ass Prof, University of California, San Diego
Allocation: Randomized | Masking: None
Other Study IDs: RCT 131309
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Hemodialysis Catheter-related Bacteremia
MeSH Terms: interventions — Tigecycline; Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antibiotic Lock Solution (Experimental)
  Interventions: Drug: tigecycline, N-acetylcysteine, heparin combination
- Guide-wire Exchange (Active Comparator)
  Interventions: Device: guide-wire exchange

INTERVENTIONS:
Drug: tigecycline, N-acetylcysteine, heparin combination
  Arms: Antibiotic Lock Solution
Device: guide-wire exchange
  Arms: Guide-wire Exchange

SUMMARY:
Patients who undergo hemodialysis via a tunneled catheter often develop bloodstream infections that arise from the catheter. There are several management options for treatment of such an infection, though the best option is not clearly delineated. Standard of care options include exchanging the catheter for a new one over a guide-wire and instilling a high concentration of an antibiotic directly into the catheter lumen. The investigators are planning to treat hemodialysis catheter bloodstream infections by one of two strategies: 1. Use of a novel antibiotic lock solution Or 2. Changing out the infected catheter for a new one. Both these options have comparable cure rates as shown in the medical literature. After obtaining informed consent, patients will be randomized to either treatment arm and will continue to receive all other standard medical care.

Specific Aim: To conduct a randomized clinical trial to demonstrate that the use of a novel antibiotic lock solution (consisting of N-acetylcysteine, tigecycline and heparin) is non-inferior to guide-wire exchange in the treatment of hemodialysis catheter-related bacteremia.

ELIGIBILITY:
Inclusion Criteria:

* Any adult (≥ 18 years of age) who has ESRD and a prevalent or incident tunneled hemodialysis catheter with bacteremia will be eligible for enrollment.

Exclusion Criteria:

* The following patients will be excluded: 1) patient is unable (and no guardian or legal representative is available) or unwilling to provide informed consent, 2) patient is allergic to NAC, tigecycline, minocycline, or heparin, 3) patient has evidence of a complicated bacteremia such as endocarditis, septic thrombophlebitis, septic emboli, osteomyelitis, deep seated abscess, or hypotension requiring use of vasopressors, 4) patient has evidence of an exit site infection around the catheter such as a pus pocket, purulent drainage, or erythema, 5) patient is pregnant or will become pregnant, 6) the infection is due to an organism that is resistant to tigecycline such as Candida or Pseudomonas species.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Success | 28 days
  The primary outcome is successful treatment of infection defined as clinical and microbiologic resolution of the initial bacteremia with absence of persistent or recurrent catheter-related bacteremia at day 28 (one week after end of treatment).

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego Medical Center, San Diego, California, United States

REFERENCES:
- [Background] Aslam S, Trautner BW, Ramanathan V, Darouiche RO. Pilot trial of N-acetylcysteine and tigecycline as a catheter-lock solution for treatment of hemodialysis catheter-associated bacteremia. Infect Control Hosp Epidemiol. 2008 Sep;29(9):894-7. doi: 10.1086/590192. PMID 18643743
- [Derived] Almeida BM, Moreno DH, Vasconcelos V, Cacione DG. Interventions for treating catheter-related bloodstream infections in people receiving maintenance haemodialysis. Cochrane Database Syst Rev. 2022 Apr 1;4(4):CD013554. doi: 10.1002/14651858.CD013554.pub2. PMID 35363884